CLINICAL TRIAL: NCT06861335
Title: Examination of the Effects of Pelvic Floor Muscle Exercises on Vulvovaginal, Umbilical, Uterine and Middle Cerebral Artery Blood Flow in Pregnant Women
Brief Title: Examination of the Effects of Pelvic Floor Muscle Exercises on Blood Flow in Pregnant Women
Acronym: Bloodflow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Melda Baser Secer, Lecturer PhD, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CelalBayarU11; Dokuz Eylul University (Other: Dokuz Eylul University medical school ethics committee)
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pelvic Floor Muscle Training; Pregnancy; Blood Flow Indexes
Keywords: pelvic floor muscle training, MCA, uterine artery, pregnancy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): Participants will undergo pelvic floor muscle training
  Interventions: Other: Exercise
- Control group (Other): Participants received standard prenatal care, education on pelvic floor health, general health education, and lifestyle counseling
  Interventions: Behavioral: Control

INTERVENTIONS:
Other: Exercise — For each participant included in the exercise group, an individualized pelvic floor muscle exercise program will be created based on the results of digital palpation and the PERFECT assessment system. The first exercise session will be conducted with the physiotherapist, and the participant will be provided with a home-based program. During pregnancy check-ups, the pelvic floor muscles will be re-evaluated, and the exercise program will be updated according to the new evaluation results. To monitor the home-based program, participants will be given an exercise tracking chart that they will be asked to fill out daily
  Arms: Exercise group
Behavioral: Control — Participants in the control group of our study will receive standard pregnancy care and check-ups. Within this scope, the general health status of the pregnant women will be evaluated during routine antenatal follow-up visits, check-ups appropriate to their gestational weeks will be performed, and necessary medical interventions will be carried out. Additionally, participants will receive detailed education about pelvic floor anatomy, the functions of the pelvic floor muscles, and the changes that occur in these muscles during pregnancy. Within the scope of general health education, information will be provided about nutrition, hygiene, exercise, and other lifestyle recommendations during pregnancy. The participants in the control group will not be given the specific pelvic floor muscle training program applied in the experimental arm of the study; they will only receive standard pregnancy care and general information
  Arms: Control group

SUMMARY:
This research will be conducted on pregnant volunteers who have applied to the Department of Obstetrics and Gynecology at Dokuz Eylul University Faculty of Medicine Hospital and undergone a comprehensive examination by an Obstetrician and Gynecologist. After these participants are informed about the content of the study, a signed informed consent form will be obtained. In the study, during mutual interviews with all participants, initial assessments will include a data recording form, digital palpation and the PERFECT system to evaluate pelvic floor muscle strength and endurance, and clitoral Doppler ultrasound to evaluate vulvovaginal blood flow. Routine pregnancy assessments will also include umbilical, uterine artery, and MCA Doppler ultrasound. Participants will be divided into two groups: exercise and control. Pregnant women in the exercise group will receive an individualized pelvic floor exercise program created by a physiotherapist (individual exercise sessions will be arranged based on data obtained from each participant's pelvic floor examination), with the first session conducted with the physiotherapist, and then they will be asked to continue this as a home program. Participants will be reassessed during their routine doctor check-ups throughout the pregnancy, and the exercise program will be updated by the physiotherapist. An exercise tracking chart will be created and given to the participants for the home program, and they will be asked to fill these out daily. Pregnant women in the control group will only receive education about the pelvic floor muscles, their functions, pelvic structure, and changes in these structures during pregnancy. Assessments will be repeated from the 2nd trimester until delivery during the participants' routine doctor check-ups. The differences between these two groups in the obtained data will be examined.

DETAILED DESCRIPTION:
This research will be conducted on pregnant women aged 18 and over, with their first pregnancy, who apply to the Department of Obstetrics and Gynecology at Dokuz Eylul University Faculty of Medicine Hospital. Participants will be informed about the purpose of the study and the assessment methods to be applied, and informed consent forms will be obtained from each participant. The demographic information of the participants will be recorded in the evaluation form.

The sociodemographic characteristics of the individuals will be evaluated through face-to-face interviews, and physical characteristics such as age (years), height (cm), weight (kg), BMI (kg/m²), and demographic data such as education level, occupation, and marital status will be recorded in the data recording form. In addition, past and family medical history, lifestyle habits, medical and surgical history, obstetric history, gynecological history, and pregnancy history will be questioned (Appendix 4). In the study, digital palpation with the PERFECT evaluation system will be used to assess pelvic floor muscle strength, and clitoral Doppler ultrasound will be used to assess vulvovaginal blood flow. Umbilical, uterine artery, and MCA blood flow will be measured by Doppler ultrasound during routine pregnancy check-ups. Assessments will be repeated three times from the 2nd trimester onwards, during the participants' regular doctor check-ups. After the first interview, participants will be randomized into exercise and control groups.

An individualized pelvic floor muscle exercise program will be created for each participant in the exercise group based on their digital palpation and PERFECT values, and will be taught in the first session with the physiotherapist, and they will be asked to do this as a home program. During the weeks they come for pregnancy check-ups, the pelvic floor muscles will be re-evaluated and the exercise program will be updated according to the new evaluation results. An exercise tracking chart will be created and given to control the home program, and participants will be asked to keep this daily and follow-up will be done. Pregnant women in the control group will not be given any exercise program and will continue their routine pregnancy follow-ups. All assessments will be repeated three times during their routine pregnancy check-ups. Separate WhatsApp groups will be created for the control and exercise groups. Reminders will be made in the exercise WhatsApp group to encourage regular exercise. Routine pregnancy information will be shared in the control WhatsApp group

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Having at least a primary school education
* Being pregnant for the first time
* Being in the 12th week of pregnancy or later
* Having a singleton pregnancy
* Having signed the informed voluntary consent form

Exclusion Criteria:

* Multiple pregnancies
* Pregnant women with pregnancy-related symptoms (hypertension, preeclampsia, gestational diabetes...)
* Pregnant women considered high-risk by an obstetrician
* Pregnant women at risk of premature birth, early delivery, or miscarriage
* Pregnant women diagnosed with neurological diseases
* Pregnant women with severe back pain (regularly unable to perform tasks)
* Pregnant women diagnosed with psychiatric diseases
* Pregnant women with severe cognitive impairment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 47 (Actual)
Dates: Start 2024-12-27 (Actual); Primary Completion 2025-04-27 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
uterine artery blood flow | The first measurement will be performed between the 20th and 24th weeks of pregnancy, the second measurement between the 25th and 28th weeks of pregnancy, and the third measurement between the 35th and 38th weeks of pregnancy.
  Uterine artery Doppler measurement is an important non-invasive method used to evaluate uteroplacental blood flow during pregnancy. This measurement is performed bilaterally from the region where the uterine arteries cross the external iliac arteries, using an abdominal ultrasonography probe. The 2nd or 3rd trimesters are generally preferred for measurement.
  Procedure:
  Patient Position: The pregnant woman is placed comfortably in a supine position. The abdominal area is exposed to allow easy movement of the probe.
  Equipment: A Doppler ultrasonography device (e.g., Voluson E8, GE Healthcare) and an abdominal probe with an appropriate frequency are used.
  Probe Placement: First, the probe is placed in the sagittal plane at the level of the internal cervical os. From this point, the probe is moved slightly towards the region where the uterine arteries cross the external iliac arteries.
  Color Doppler: Color Doppler mode is used to visually identify the uterine arteries. Color Doppler dis
umbilical artery blood flow | The first measurement will be performed between the 20th and 24th weeks of pregnancy, the second measurement between the 25th and 28th weeks of pregnancy, and the third measurement between the 35th and 38th weeks of pregnancy.
  Umbilical artery waveform patterns can be obtained from either of the two arteries in the umbilical cord using color Doppler and pulsed Doppler. The angle of the probe to the vessel should be below 60°. It is important to perform the measurements from the freest point where the umbilical vessels are not compressed. The umbilical artery waveform shows systolic (heart contraction) and diastolic (heart relaxation) flow. Pulsatility index (PI) are calculated.
middle cerebral artery blood flow | The first measurement will be performed between the 20th and 24th weeks of pregnancy, the second measurement between the 25th and 28th weeks of pregnancy, and the third measurement between the 35th and 38th weeks of pregnancy.
  To obtain an ideal waveform in the middle cerebral artery (MCA) measurement, the Circle of Willis and the proximal MCA color flow mapping just caudal to the transthalamic plane will be visualized. The probe will then be placed at the proximal third of the MCA, close to its origin from the internal carotid artery, keeping the insonation angle as close to 0° as possible [48]. Doppler indices will be calculated by obtaining 3 consecutive waveforms. Middle cerebral artery Doppler measurement is routinely performed in pregnancy examinations to assess pregnancy complications. Measurements will be performed by an obstetrician during routine pregnancy check-ups.
vulvovaginal blood flow | The first measurement will be performed between the 20th and 24th weeks of pregnancy, the second measurement between the 25th and 28th weeks of pregnancy, and the third measurement between the 35th and 38th weeks of pregnancy.
  Doppler ultrasonography (Voluson E8, GE Healthcare, Salzburg, Austria) will be used to identify the dorsal clitoral artery, sampled from the outer surface of the clitoral body, in a longitudinal plane. With the same longitudinal approach, the terminal branch of the posterior labial artery (a branch of the internal pudendal artery) will be visualized posterolaterally to the labia majora (approximately 2 cm away from the clitoral hood). For both the clitoral and labial arteries, the insonation angle will always be adjusted (<40°) to obtain maximum color intensity. Once adequate signals are obtained, blood flow velocity waveforms will be recorded by placing the spectral Doppler gate along the vessel and activating the pulsed Doppler mode. The Pulsatility Index (PI), defined as the difference between peak systolic and end-diastolic flow divided by the mean maximum flow velocity, will be calculated electronically by the machine.
pelvic floor muscle function | The first measurement will be performed between the 20th and 24th weeks of pregnancy, the second measurement between the 25th and 28th weeks of pregnancy, and the third measurement between the 35th and 38th weeks of pregnancy.
  The patient is asked to squeeze one or two fingers placed inside the vagina, and the strength of the contraction felt around the fingers is graded according to various scales. Physiotherapists most commonly use the Modified Oxford Grading Scale developed by Laycock in clinical practice to measure pelvic floor muscle strength. In 2001, the PERFECT Scale was developed by Laycock. The PERFECT Scale allows for the evaluation of the strength (P).
pelvic floor muscle function | The first measurement will be performed between the 20th and 24th weeks of pregnancy, the second measurement between the 25th and 28th weeks of pregnancy, and the third measurement between the 35th and 38th weeks of pregnancy.
  The patient is asked to squeeze one or two fingers placed inside the vagina, and the strength of the contraction felt around the fingers is graded according to various scales. Physiotherapists most commonly use the Modified Oxford Grading Scale developed by Laycock in clinical practice to measure pelvic floor muscle strength. In 2001, the PERFECT Scale was developed by Laycock. The PERFECT Scale allows for the evaluation of the endurance (E).
pelvic floor muscle function | The first measurement will be performed between the 20th and 24th weeks of pregnancy, the second measurement between the 25th and 28th weeks of pregnancy, and the third measurement between the 35th and 38th weeks of pregnancy.
  The patient is asked to squeeze one or two fingers placed inside the vagina, and the strength of the contraction felt around the fingers is graded according to various scales. Physiotherapists most commonly use the Modified Oxford Grading Scale developed by Laycock in clinical practice to measure pelvic floor muscle strength. In 2001, the PERFECT Scale was developed by Laycock. The PERFECT Scale allows for the evaluation fast-twitch muscle fiber performance (F).

CONTACTS AND LOCATIONS:
Overall Officials: Özge Çeliker Tosun, professor, Principal Investigator — Dokuz Eylul University
Locations (1):
- Manisa Celal Bayar Univercity, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
all IPD collected throughout the trial, only IPD used in the results publication

REFERENCES:
- [Derived] Baser Secer M, Ci̇cek Guvendi̇k S, Celiker Tosun O, Yavuz O, Kurt S, Tosun G, Basol Goksuluk M. The hidden power in the miracle of pregnancy: the effect of pelvic floor muscle training on fetal and fetal-maternal blood circulation and pelvic floor muscles during pregnancy, a randomized controlled trial. BMC Pregnancy Childbirth. 2025 Nov 19;25(1):1241. doi: 10.1186/s12884-025-08412-3. PMID 41257651